CLINICAL TRIAL: NCT03974945
Title: Can Sensory Feedback Training Improve the Biomechanical and Metabolic Effects of Using Passive or Powered Lower Limb Prostheses During Walking for Veterans With Transtibial Amputations?
Brief Title: Does Walking Performance Improve When Veterans With Leg Amputations Are Given Visual Feedback?
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A2943-R
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Amputation
Keywords: Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — none retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Transtibial Amputation: The investigators will recruit participants with unilateral transtibial amputations who are at or above a K3 Medicare functional classification level (MFCL), and 18-60 years old. A K3 MFCL means that a person has the ability or potential for ambulation with variable cadence. A person at K3 MFCL is a typical community ambulator who has the ability to traverse most environmental barriers and may have vocational, therapeutic or exercise activity that demands prosthetic use beyond simple locomotion.
  Interventions: Device: Passive-elastic prosthetic foot; Device: Powered ankle-foot prosthesis

INTERVENTIONS:
Device: Passive-elastic prosthetic foot — The investigators will measure the biomechanics (motion, forces, and muscle activity) and metabolic rates while subjects walk using their own passive-elastic prosthesis with and without visual feedback of peak propulsive force targets.
Device: Powered ankle-foot prosthesis — The investigators will measure the biomechanics (motion, forces, and muscle activity) and metabolic rates while subjects walk using a battery-powered ankle-foot prosthesis with and without visual feedback of peak propulsive force targets.

SUMMARY:
Previous studies suggest that Veterans with below the knee amputation using passive-elastic or powered prostheses have impaired physical function, which could increase the risk of osteoarthritis, leg/back pain, and diabetes/obesity. Utilization of rehabilitation strategies/techniques such as real-time visual feedback training could restore physical function, increase physical activity, and reduce injury risk. The investigators will systematically determine the effects of using real-time visual feedback training of peak propulsive (push-off) force during walking while Veterans with below the knee amputations use a passive-elastic and battery-powered prosthesis. Similar to previous studies of non-amputee older (>65 years) and post-stroke adults, use of real-time visual feedback training of propulsive force will likely improve walking function in Veterans with amputations. Such training presents a promising rehabilitation strategy that could reduce comorbidities, while improving quality of life, comfort, and physical function, and advancing rehabilitation research and prosthetic development.

DETAILED DESCRIPTION:
Due to the functional impairments caused by a lower limb amputation, it is essential to determine the benefits of rehabilitation strategies such as real-time visual feedback training. Such training could allow Veterans with transtibial amputations (TTAs) to better utilize their prostheses and regain the greatest possible level of function. It is not clear how much the prosthetic device (passive-elastic prosthetic foot versus battery-powered ankle-foot prosthesis) and/or the user's response to the prosthesis contribute to the biomechanical and metabolic effects of using these prostheses during walking. Better use of a prosthesis due to targeted real-time visual feedback training could enhance rehabilitation, improve function and reduce asymmetric biomechanics, which in turn could reduce common comorbidities such as osteoarthritis, leg and back pain, and indirectly, diabetes in Veterans with TTAs. The purpose of the proposed project is to systematically establish the metabolic and biomechanical effects of targeted real-time visual feedback training of peak propulsive ground reaction force (GRF) on the biomechanics, metabolic costs, and muscle activity of Veterans with TTAs using their own passive-elastic prosthetic foot and a battery-powered ankle-foot prosthesis. The results of the investigators' research could enhance the use of prosthetic technology to improve the rehabilitation and function of Veterans with lower limb amputations.

Previous studies suggest that use of passive-elastic and/or powered ankle-foot prostheses may not optimize the function of Veterans with TTAs during walking. Targeted, real-time visual feedback training of peak propulsive ground reaction forces increased propulsion and improved walking function in older (>65 years) and post-stroke adults, who typically have impaired ankle power. To the investigators' knowledge, no research has addressed how visual feedback of peak propulsive force affects the use of passive-elastic or powered ankle-foot prostheses by people with TTAs. In the proposed research, the investigators will determine the underlying metabolic costs, biomechanics, stability, and muscle activity resulting from targeted real-time visual feedback training of peak propulsive force to identify how Veterans with a TTA benefit from more effective use of a passive-elastic prosthesis and/or a battery-powered ankle-foot prosthesis and to determine if the addition of mechanical power provided by a battery-powered ankle-foot prosthesis can further enhance the function of Veterans with unilateral TTAs during walking. 30 Veterans with unilateral TTAs will use their own passive-elastic prosthesis both with and without visual feedback training during level-ground walking, while the investigators measure their metabolic costs and biomechanics. Then, they will use a powered ankle-foot prosthesis (emPOWER, BiONX, Ottobock) both with and without visual feedback training during level-ground walking, while the investigators measure their metabolic costs and biomechanics. With each prosthesis, subjects will walk at 1.25 m/s on a dual-belt force-measuring treadmill 1) with no visual feedback, and then with real-time visual feedback of: 2) peak propulsive force from the "no feedback" condition, 3) +20% greater peak propulsive force, and 4) +40% greater peak propulsive force. During these visual feedback trials, the investigators will ask subjects to match the peak propulsive force displayed on a computer screen with their affected leg. The investigators will also ask subjects to: 5) match symmetric visual feedback of the peak propulsive force from both legs. The investigators will determine if Veterans with TTAs utilizing real-time visual feedback training of peak propulsive force can improve metabolic costs, biomechanical symmetry, and dynamic stability/balance, while using their own passive-elastic prosthesis or a powered ankle-foot prosthesis. The investigators will also establish if Veterans with TTAs can retain the metabolic and biomechanical benefits elicited by real-time visual feedback training once that feedback is removed. Results from the proposed project will be used to inform rehabilitation strategies and prosthetic design, which could ultimately improve health, maximize function, and improve quality of life for Veterans with TTAs.

ELIGIBILITY:
Inclusion Criteria:

* One amputation below the knee
* At least 1 year of experience using a prosthesis
* No current problems with the prosthesis or residual limb
* At or above a K3 Medicare Functional Classification Level

Exclusion Criteria:

* Poor general health
* Difficulty with mobility
* Problems with balance or dizziness
* Current serious musculoskeletal injury besides that associated with an amputation
* Cardiovascular, pulmonary, or neurological disease or disorder

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit 30 subjects with unilateral transtibial amputations from the VA Jewell Clinic, locally, and nationally.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alena Grabowski, PhD BA, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Transtibial Amputation
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Transtibial Amputation
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Affected Leg Peak Propulsive Horizontal Ground Reaction Force
Description: The investigators measured peak propulsive horizontal ground reaction force (hGRFpeak) from the affected leg while participants with a transtibial amputation walked at 1.25 m/s for 18 trials that were 5 minutes each over 3 separate days using an elastic energy storage and return (ESAR) and stance-phase powered ankle-foot (BiOM) prosthesis. During the first trial we measured their baseline hGRFpeak and then for the subsequent trials we provided a trial with visual feedback (FB) targets of hGRFpeak relative to their baseline (BL) trial using a monitor placed at eye level as well as VF of symmetric (Sym) targets of hGRFpeak from both legs and then removed the visual feedback during a retention (RT) trial that immediately followed the VF trial. The order of trials was randomized and included targets of 0, +20, and +40% of baseline hGRFpeak as well as a Sym target of hGRFpeak. Thus, participants performed 9 trials per prosthesis.
Time Frame: 18 trials that are 5 minutes in length
Measure: Mean (Standard Deviation); unit: proportion of body weight
Groups:
- ESAR - BL; BiOM - BL: Baseline no feedback
- ESAR - 0FB; BiOM - 0FB: Baseline feedback
- ESAR - 0RT; BiOM - 0RT: Baseline retention
- ESAR - 20FB; BiOM - 20FB: +20% feedback
- ESAR - 20RT; BiOM - 20RT: +20% retention
- ESAR - 40FB; BiOM - 40FB: +40% feedback
- ESAR - 40RT; BiOM - 40RT: +40% retention
- ESAR - SymFB; BiOM - SymFB: Symmetry feedback
- ESAR - SymRT; BiOM - SymRT: Symmetry retention
Arm/Group | ESAR - BL | ESAR - 0FB | ESAR - 0RT | ESAR - 20FB | ESAR - 20RT | ESAR - 40FB | ESAR - 40RT | ESAR - SymFB | ESAR - SymRT | BiOM - BL | BiOM - 0FB | BiOM - 0RT | BiOM - 20FB | BiOM - 20RT | BiOM - 40FB | BiOM - 40RT | BiOM - SymFB | BiOM - SymRT
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
proportion of body weight | 0.151 (0.022) | 0.145 (0.019) | 0.166 (0.021) | 0.150 (0.022) | 0.175 (0.020) | 0.147 (0.018) | 0.145 (0.022) | 0.171 (0.031) | 0.146 (0.022) | 0.169 (0.011) | 0.160 (0.011) | 0.178 (0.021) | 0.161 (0.011) | 0.186 (0.020) | 0.166 (0.014) | 0.157 (0.018) | 0.174 (0.019) | 0.172 (0.024)

2. Primary Outcome: Net Metabolic Power
Description: The investigators measured net metabolic power while participants with a transtibial amputation walked at 1.25 m/s for 18 trials that were 5 minutes each over 3 separate days using an elastic energy storage and return (ESAR) and stance-phase powered ankle-foot (BiOM) prosthesis. During the first trial we measured their baseline peak propulsive horizontal ground reaction force (hGRFpeak) from the affected leg and then for the subsequent trials we provided a trial with visual feedback (FB) targets of hGRFpeak relative to their baseline (BL) trial using a monitor placed at eye level as well as VF of symmetric (Sym) targets of hGRFpeak from both legs and then removed the visual feedback during a retention (RT) trial that immediately followed the VF trial. The order of trials was randomized and included targets of 0, +20, and +40% of baseline hGRFpeak as well as a Sym target of hGRFpeak. Thus, participants performed 9 trials per prosthesis.
Time Frame: 18 trials that are 5 minutes in length
Measure: Mean (Standard Deviation); unit: Watts per kg
Arm/Group | ESAR - BL | ESAR - 0FB | ESAR - 0RT | ESAR - 20FB | ESAR - 20RT | ESAR - 40FB | ESAR - 40RT | ESAR - SymFB | ESAR - SymRT | BiOM - BL | BiOM - 0FB | BiOM - 0RT | BiOM - 20FB | BiOM - 20RT | BiOM - 40FB | BiOM - 40RT | BiOM - SymFB | BiOM - SymRT
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Watts per kg | 2.967 (0.345) | 3.141 (0.275) | 3.020 (0.230) | 3.338 (0.422) | 3.124 (0.316) | 3.478 (0.488) | 3.168 (0.409) | 3.330 (0.554) | 3.062 (0.317) | 2.852 (0.413) | 2.979 (0.436) | 2.938 (0.425) | 3.268 (0.561) | 3.022 (0.473) | 3.314 (0.540) | 3.013 (0.418) | 2.974 (0.539) | 2.862 (0.399)

3. Primary Outcome: Trailing Affected Leg Positive Work
Description: The investigators measured ground reaction forces and calculated individual leg work during step to step transitions while participants with a transtibial amputation walked at 1.25 m/s for 18 trials that were 5 minutes each over 3 separate days using an elastic energy storage and return (ESAR) and stance-phase powered ankle-foot (BiOM) prosthesis. During the first trial we measured their baseline peak propulsive horizontal ground reaction force (hGRFpeak) from the affected leg and then for the subsequent trials we provided a trial with visual feedback (FB) targets of hGRFpeak relative to their baseline (BL) trial using a monitor placed at eye level as well as VF of symmetric (Sym) targets of hGRFpeak from both legs and then removed the visual feedback during a retention (RT) trial that immediately followed the VF trial. The order of trials was randomized and included targets of 0, +20, and +40% of baseline hGRFpeak as well as a Sym target of hGRFpeak.
Time Frame: 18 trials that are 5 minutes in length
Measure: Mean (Standard Deviation); unit: Joules
Arm/Group | ESAR - BL | ESAR - 0FB | ESAR - 0RT | ESAR - 20FB | ESAR - 20RT | ESAR - 40FB | ESAR - 40RT | ESAR - SymFB | ESAR - SymRT | BiOM - BL | BiOM - 0FB | BiOM - 0RT | BiOM - 20FB | BiOM - 20RT | BiOM - 40FB | BiOM - 40RT | BiOM - SymFB | BiOM - SymRT
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Joules | 9.859 (3.392) | 10.321 (4.325) | 10.773 (4.326) | 10.212 (4.419) | 11.203 (4.652) | 10.319 (4.463) | 9.592 (4.212) | 11.384 (3.941) | 10.410 (4.642) | 14.624 (5.800) | 14.108 (4.835) | 15.211 (6.363) | 13.597 (5.413) | 15.274 (6.466) | 14.071 (4.450) | 12.818 (4.203) | 14.730 (6.242) | 15.078 (5.575)

4. Primary Outcome: Leading Unaffected Leg Negative Work
Description: as for outcome 3
Time Frame: 18 trials that are 5 minutes in length
Measure: Mean (Standard Deviation); unit: Joules
Arm/Group | ESAR - BL | ESAR - 0FB | ESAR - 0RT | ESAR - 20FB | ESAR - 20RT | ESAR - 40FB | ESAR - 40RT | ESAR - SymFB | ESAR - SymRT | BiOM - BL | BiOM - 0FB | BiOM - 0RT | BiOM - 20FB | BiOM - 20RT | BiOM - 40FB | BiOM - 40RT | BiOM - SymFB | BiOM - SymRT
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Joules | -15.373 (4.191) | -14.438 (4.394) | -15.981 (6.225) | -14.363 (4.590) | -17.781 (7.167) | -14.018 (5.195) | -14.389 (4.451) | -15.350 (6.056) | -14.223 (5.517) | -15.781 (6.674) | -15.011 (6.284) | -17.975 (5.403) | -14.713 (5.840) | -18.475 (7.963) | -16.032 (6.839) | -15.507 (5.169) | -15.755 (6.950) | -14.918 (5.957)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of the study, which was ~4 years, 9 months. Each participant was assessed in relation to their first session through their completion of the study, which was up to a month after the first session.
Arm/Group | Participants With Transtibial Amputation
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT03974945/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT03974945/ICF_000.pdf